CLINICAL TRIAL: NCT07039097
Title: A Multicenter, Prospective, Randomized, Controlled Clinical Study on the Effect of Hysteroscopic Uterine Septum Resection on the Natural Pregnancy Outcomes in Patients With Non-recurrent Spontaneous Abortion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other); Peking Union Medical College Hospital (Other); Maternal and Child Health Hospital of Hubei Province (Other); Beijing Tiantan Hospital (Other); Anhui Provincial Hospital (Other Government); Beijing Fuxing Hospital (Unknown); Tongji Hospital (Other); The First People's Hospital of Yunnan (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Southwest Hospital, China (Other); The First Hospital of Jilin University (Other); Tianjin Medical University General Hospital (Other); Xijing Hospital (Other); Hospital for Reproductive Medicine Affiliated to Shandong University (Unknown); Guangzhou First People's Hospital (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xy3-TCRS-NP
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Infertility and Miscarriage
Keywords: transcervical resection of septum; Natural Pregnancy
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical group (Experimental): Undergoing Transcervical resection of septum
  Interventions: Procedure: Transcervical resection of septum
- Control group (No Intervention): Routine preconception counseling and observation without hysteroscopic septectomy

INTERVENTIONS:
Procedure: Transcervical resection of septum — Transcervical resection of septum (TCRS) is divided into two categories: one is plasma hysteroscopic electrosurgical resection (actually TCIS), which uniformly uses a 7mm external diameter hysteroscopic electrosurgical resectoscope to reduce the difficulty of cervical dilation; the other is micro (5 or 7Fr) hysteroscopic cold knife incision, equipped with a 5Fr bipolar electrocoagulation stick for electrocoagulation and hemostasis.
  Arms: Surgical group

SUMMARY:
The study aims to compare the effects of transcervical resection of septa (TCRS) and expectant management on the natural pregnancy outcomes of patients with septate uterus without recurrent abortion, also covering the treatment of other infertility factors in infertile patients who aim at natural conception. The research attempts to answer whether TCRS can improve the live birth rate, pregnancy rate and pregnancy outcomes for septate uterus patients planning natural pregnancy, so as to provide evidence-based medical evidence for the selection of clinical treatment methods for such patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) The patient meets the 2024 ASRM diagnostic criteria for uterine septate after three-dimensional color Doppler ultrasound examination; (2) The patient may have never been pregnant, or may have a history of live birth, one biochemical pregnancy, or one fetal arrest. The patient may also be an infertile patient who wishes to conceive naturally, such as a patient with hydrosalpinx and laparoscopic stoma, or a patient whose infertility factors can be treated; (3) The patient is between 20 and 40 years old; (4) The patient plans to try to conceive naturally to achieve the desire to have a baby; (5) The patient has normal ovarian reserve function (AMH>1.1ng/ml, FSH<12U/L on the 2nd to 5th day of menstruation); (6) The male's semen is generally normal; (7) The patient signs the informed consent form and is able to accept and adhere to treatment and follow-up. Patients in the control group can undergo hysteroscopy or hystero-laparoscopy to treat other problems, but septal resection is not performed.

Exclusion Criteria:

* (1) Recurrent miscarriage; (2) Patients with intramural uterine myoma larger than 3 cm, moderate to severe intrauterine adhesions; (3) Uncontrolled endocrine disorders, such as abnormal thyroid function (FT3, FT4 abnormal), hyperprolactinemia (greater than 2 times the upper limit of normal), uncontrolled endometrial hyperplasia, EIN or malignant lesions, acute inflammation of the reproductive system, coagulation dysfunction, etc.; if combined with endometrial polyps or submucosal myoma, patients can still be included in the group after resection; (4) Patients with adenomyosis (uterine body>50 days of pregnancy), chocolate cysts with a diameter of>4 cm, or severe dysmenorrhea and clear DIE lesions (diameter>1 cm) can be palpated during gynecological triple examination; (5) Untreated bilateral hydrosalpinx or obstruction; (6) Other important organ diseases and other surgical contraindications or relative contraindications. Other situations that are not suitable for assisted reproductive treatment. Those who have participated in other clinical research (within the past three months); (7) Those who are assessed to need IVF (e.g., those whose fallopian tubes cannot be cleared, or whose ovulation dysfunction cannot be treated with medication, etc.).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 418 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
live birth rate | within 12 months after initiating embryo transfer
  Follow-up was conducted for 12 months after the surgery or treatment course to record the IVF/ICSI reproductive outcomes within 12 months after the initiation of embryo transfer into the cycle.

SECONDARY OUTCOMES:
Adverse outcome rate | within 12 months after initiating embryo transfer in both groups
  Pregnancy rate and cumulative pregnancy rate, miscarriage rate and cumulative miscarriage rate, preterm birth rate.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT07039097/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT07039097/ICF_001.pdf